CLINICAL TRIAL: NCT07121699
Title: The Role of Left Ventricular Outflow Tract (LVOT) Velocity-time Integral (VTI) and Respiratory Variability at Peak Rate (Vpeak) in Predicting Hypotension After General Anesthesia Induction
Acronym: LVOT-VTI-hypot
Status: Not yet recruiting | Type: Observational
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, ferdi gülaştı, asst. prof.dr, Aydin Adnan Menderes University
Other Study IDs: 2025-08
Record Dates: First submitted 2025-08-07; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Hypotension on Induction
Keywords: respiratory variability in peak velocity (Vpeak); left ventricular outflow tract (LVOT) velocity-time integral (VTI); general anesthesia; hypotension
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- with hypotension: Patients with a 30% decrease in SBP from baseline and a decrease in MAP below 65 mmHg in the first 10 minutes after anesthesia induction will be considered to have hypotension.
  Interventions: Drug: Inotrope
- none hypotension: Patients with a 30% decrease in SBP from baseline and a decrease in MAP below 65 mmHg in the first 10 minutes after anesthesia induction will be considered to have hypotension.

INTERVENTIONS:
Drug: Inotrope — Hypotensive attacks with MAP below 55 mmHg or prolonged duration (2 minutes or more) will be treated with ephedrine 0.1 mg/kg.
  Groups: with hypotension

SUMMARY:
Preoperatively, patients will undergo transthoracic echocardiography measurements approximately 15-30 minutes before induction. TTE will be performed on all patients by an experienced observer; the echocardiography device will be equipped with an S4-2 transducer (4-2 MHz frequency range) in the left lateral decubitus position.

VTI and Vpeak values of the LVOT were measured from manually drawn contours using pulsatile wave Doppler technique in the apical five-chamber view. The Doppler beam was aligned with the aortic blood flow, and the signal was captured at an appropriate angle (<20°).

The maximum (VTImax) and minimum (VTImin) VTI, as well as the maximum (Vpeakmax) and minimum (Vpeakmin) Vpeak values, were determined over three respiratory cycles. ΔVTI was calculated with the following formula:

ΔVTI = [2 × (VTImax - VTImin) / (VTImax + VTImin)] × 100%.

ΔVpeak was calculated with the following formula:

ΔVpeak = [2 × (Vpeakmax - Vpeakmin) / (Vpeakmax + Vpeakmin)] × 100%. These parameters were analyzed to evaluate the hemodynamic status of patients and estimate fluid responsiveness.

Patients with a 30% decrease from baseline in SBP and a decrease in MAP below 60 mmHg in the first 10 minutes after anesthesia induction were considered to have hypotension. Patients were divided into two groups: "with" and "without" hypotension.

DETAILED DESCRIPTION:
The study is planned to be conducted for one year after receiving approval from the non-invasive clinical research ethics committee. Documentation of eligibility and consent will be confirmed at the preoperative visit. During this visit, patients will provide demographic and past medical information, including medication use.

Preoperative transthoracic echocardiography measurements will be performed on all patients 15-30 minutes before induction. TTE will be performed by an experienced observer; the echocardiography device is equipped with an S4-2 transducer (4-2 MHz frequency range) in the left lateral decubitus position. LV Ejection Fraction (EF) measurements will be evaluated in the parasternal long-axis view. ΔVTI and ΔVpeak, and LVOT will be recorded.

Patients will be positioned supine, and the Inferior Vena Cava (IVC) will be imaged through the subxiphoid window. The cursor will be placed 1 cm distal to the hepatic vein IVC entry point, and the IVC diameter will be monitored in M-Mode for 30 seconds. The measurement will be taken at the site where the inferior vena cava diameter is measured during inspiration (IVCins) and expiration (IVCexp) while the patient is breathing normally. Inferior Vena Cava Collapse Ratio (IVC-CI) will be calculated using the formula IVC-CI = (IVCexp - IVCins) / IVCexp.

Intraoperative The patient will be administered the clinic's routine anesthesia protocol. Anesthesia will not be interfered with.

Our clinic's routine anesthesia protocol includes: fentanyl 1μg/kg IV, propofol 1.5 to 2.5 mg/kg IV, lidocaine 1 mg/kg IV, and rocuronium 0.6 mg/kg IV. Sevoflurane 2% is initiated after intubation. Perioperative mean blood pressure will be targeted above 65 mmHg. Hypotension below 65 mmHg MAP will be recorded intraoperatively and postoperatively.

The first post-induction measurement will be taken before tracheal intubation. Baseline hemodynamic parameters and non-invasive and/or hemodynamic values will be recorded every two minutes after induction until the surgical incision. Patients will then undergo urinary catheterization and surgical field preparation. MAP below 55 mmHg or prolonged hypotensive episodes (2 minutes or more) will be treated with ephedrine 0.1 mg/kg. Patients with a 30% decrease from baseline in SBP and a MAP below 65 mmHg in the first 10 minutes after anesthesia induction will be considered hypotension. Patients will be divided into two groups: "with" and "without" hypotension.

E-MEASUREMENTS Demographic data to be obtained will include recording height (cm), weight (kg), age (years), gender, (ASA) physical status, and the specific procedure type. Patients will be questioned about tobacco, alcohol, and drug use. They will also be asked about their medical history, including lung disease, kidney disease, diabetes mellitus, neurological disease, chronic pain conditions, previous surgery or stent placement, and medications. Current preoperative laboratory tests and medication list will be recorded.

The amount of intraoperative bleeding, the amount of blood and blood product transfusions, and the duration of surgery will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years
* ASA Physical Status 1-3;
* Patients scheduled for general anesthesia

Exclusion Criteria:

1. Patient is pregnant
2. Post-cardiac surgery
3. Severe pulmonary hypertension
4. Severe valvular disease
5. Hypertrophic or dilated cardiomyopathy
6. Presence of acute myocardial infarction
7. Patients with severe visual or hearing impairment/impairment
8. ASA physical status IV or V
9. Ischemic heart disease, conduction disturbance
10. History of long-term use of certain medications (β-blockers, angiotensin-converting enzyme inhibitors, analgesics, sedatives, or tricyclic antidepressants)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will be conducted on hemodynamically stable patients aged between 18 and 75 years, with an American Society of Anesthesiologists (ASA) physical status classification of I-III, who are scheduled for elective surgery and will undergo general anesthesia.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-08-20 (Estimated); Primary Completion 2025-08-20 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
lvot-vtı | 1 hour
  The relationship between hypotension following induction of general anesthesia and respiratory variability in left ventricular outflow tract VTI peak velocity (Vpeak variability).

SECONDARY OUTCOMES:
lv echo | 1 hour
  The relationship between hypotension following induction of general anesthesia and left ventricular function parameters measured by transthoracic echocardiography (TTE).